CLINICAL TRIAL: NCT01276756
Title: Randomized Study for the Assessment of Nitazoxanide in the Treatment of Chronic Hepatitis C Genotype 4
Brief Title: Efficacy of Nitazoxanide in the Treatment of Chronic Hepatitis C Virus (HCV)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Egyptian Railway Hospital (Other)
Responsible Party: Principal Investigator, Hany Shehab, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAIL001
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Hepatitis c
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; nitazoxanide; Ribavirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care (Active Comparator): Group A: comprises 50 treatment-naive chronic hepatitis c patients who will receive the standard of care treatment: peginterferon Alfa 2a 160 ug once weekly and weight-based ribavirin 1000 or 1200 mg/day (based on body weight < 75 kg or ≥ 75 kg, respectively) in divided doses for 48 weeks.
  Interventions: Drug: Pegylated interferon alfa-2a; Drug: Ribavirin
- Triple therapy (Experimental): Group B: comprises 50 treatment-naive chronic HCV patients who will receive oral Nitazoxanide 500 mg twice daily for 4 weeks (lead-in phase) followed by triple therapy, nitazoxanide 500 mg twice daily plus peginterferon alfa-2a (160ug once weekly) and weight-based ribavirin 1000-1200 mg daily (based on body weight < 75 kg or ≥ 75 kg, respectively) in divided doses for 48 weeks.
  Interventions: Drug: Pegylated interferon alfa-2a; Drug: Nitazoxanide; Drug: Ribavirin

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a — Pegylated interferon 160ug once weekly 48 weeks
  Other Names: Reiferon retard
Drug: Nitazoxanide — Nitazoxanide 500mg twice daily 4 weeks lead-in followed by triple therapy 48 weeks
  Other Names: Xerovirin-C
  Arms: Triple therapy
Drug: Ribavirin — Ribavirin (> 75kg:1200 mg, <75kg:1000mg daily)48 weeks

SUMMARY:
Chronic hepatitis C has become an endemic disease in Egypt with a rising prevalence (genotype 4), worldwide it also poses a significant health burden. To date standard of care treatment (pegylated interferon and ribavirin) give modest results with a sustained virological response (SVR) of about 50%. Several pharmaceutical and herbal agents have been used with an aim to improve current results. Recent reports have suggested an increased SVR with the addition of Nitazoxanide to standard of care. The results are preliminary and need to be confirmed. This is a randomized trial to assess the efficacy of nitazoxanide added to standard of care compared to standard of care alone.

ELIGIBILITY:
Inclusion Criteria:

* Adult (male or female), 18 to 65 years of age, with chronic HCV infection
* BMI < 35
* Liver biopsy showing chronic hepatitis with significant fibrosis using Ishak scoring system
* Compensated liver disease; serum bilirubin < 1.5 mg/dl, INR (international normalized ratio) no more than 1.5, serum albumin > 3.4, platelet count > 75,000 mm, and no evidence of hepatic decompensation (hepatic encephalopathy or ascites)
* Acceptable hematological and biochemical indices (hemoglobin 13g/dl for men and 12 g/dl for women; neutrophil count 1500/mm3 or more and serum creatinine < 1.5 mg/dl
* Patients must be serum hepatitis B surface antigen (HBsAg) negative
* Negative Antinuclear Antibodies (ANA) or titer of < 1:160
* Serum positive for anti-HCV antibodies and HCV-RNA
* Abdominal Ultrasound obtained within 3 months prior to entry in the study
* Electrocardiogram for men aged > 40 years and for women aged > 50 years
* Normal fundus examination
* Ensure strict measures to avoid conception for both male and female participants by using a proper contraception measure all throughout the course of treatment and six months later
* Female patients must not breast feed during therapy

Exclusion Criteria:

* Patients who previously received interferon
* HgbA1c > 7.5 (glycoslylated haemoglobin)or history of diabetes mellitus
* BMI > 34
* Women who are pregnant or breast-feeding
* Males whose female partners are either pregnant or of child-bearing potential or not using birth control and are sexually active
* Other causes of liver disease including autoimmune hepatitis
* Transplant recipients receiving immune suppression therapy
* Screening tests positive for anti-HAV IgM Ab, HBsAg, anti-HBc IgM Ab or anti-HIV Ab
* Decompensated cirrhosis, history of variceal bleeding, ascites, hepatic encephalopathy, CTP score > 6 (Child-Turcot-Pugh) or MELD score > 8
* Absolute neutrophil count < 1500 cells/mm3; platelet count < 135,000 cells/mm3; hemoglobin < 12 g/dL for women and < 13 g/dL for men; or serum creatinine concentration ≥ 1.5 times ULN (upper limit of normal)
* Hypothyroidism or hyperthyroidism not effectively treated with medication
* Alcohol consumption of > 40 grams per day or an alcohol use pattern that will interfere with the study
* History or other clinical evidence of significant or unstable cardiac disease
* History or other clinical evidence of chronic pulmonary disease associated with functional impairment
* Serious or severe bacterial infection(s)
* History of severe or uncontrolled psychiatric disease, including severe depression, history of suicidal ideation, suicidal attempts or psychosis requiring medication and/or hospitalization
* History of uncontrolled severe seizure disorder
* History of immunologically mediated disease requiring more than intermittent anti-inflammatory medications for management or that requires frequent or prolonged use of corticosteroids
* Patients with clinically significant retinal abnormalities
* History of hypersensitivity or intolerance to nitazoxanide or any of the excipients comprising the nitazoxanide tablets, peginterferon alfa-2a injectable solution or ribavirin tablets

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hany M Shehab, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Shehab HM, Elbaz TM, Deraz DM. Nitazoxanide plus pegylated interferon and ribavirin in the treatment of genotype 4 chronic hepatitis C, a randomized controlled trial. Liver Int. 2014 Feb;34(2):259-65. doi: 10.1111/liv.12267. Epub 2013 Jul 24. PMID 23890273

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Triple Therapy
Started | 50 | 50
Completed | 45 | 48
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Triple Therapy | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.46 (6.88) | 45.42 (8.36) | 45.44 (7.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 48 | 49 | 97
Region of Enrollment [Number; unit: participants]
  Egypt | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response
Description: sustained virological response is defined as a negative HCV PCR at 180 days after the end of treatment (End of treatment being at 48 weeks for Group A, 52 weeks for Group B). For any patient who stopped treatment prematurely (e.g. due to adverse events) SVR was defined as a negative HCV PCR (polymerase chain reaction) at 180 days after the last dose of all medications (interferon, ribavirin and nitazoxanide)
Time Frame: 180 days (+- 7 days) after the end of treatment. (48 weeks for Group A, 52 weeks for Group B, or after the last dose of treatment for patients who stopped prematurely).
Population: All was intention-to-treat (ITT) analysis. Any patient who received at least one dose of interferon was included in the analyses.The only 2 dropouts (lost to follow-up) were calculated as failures.
Measure: Number; unit: participants
Arm/Group | Standard of Care | Triple Therapy
Number analyzed (Participants) | 50 | 50
participants | 24 (0.5) | 25 (0.5)

2. Secondary Outcome: Rapid Virological Response
Description: A rapid virologic response is defined as a negative HCV PCR 4 weeks after treatment
Time Frame: 28 - 33 days after start of Pegylated interferon and ribavirin
Population: Only 1 patient in "standard of care" arm and 3 patients in the "triple therapy" arm missed doing the PCR test at week 4. These patients were thus not included in this particular analysis.
Measure: Number; unit: participants
Arm/Group | Standard of Care | Triple Therapy
Number analyzed (Participants) | 49 | 47
participants | 30 | 25

3. Secondary Outcome: Early Virological Response
Description: A complete early virologic response is defined as a negative HCV PCR 90 days after the start of pegylated interferon.
  A partial early virologic response is defined as a decrease of 2 or more log in HCV PCR at 90 days after the start of pegylated interferon
Time Frame: 90 ± 7 days from the start of pegylated interferon and ribavirin
Population: ITT. Any patient who received at least one dose of interferon was included in the analyses.
Measure: Number; unit: participants
Arm/Group | Standard of Care | Triple Therapy
Number analyzed (Participants) | 50 | 50
participants
  Complete early virologic response | 35 | 36
  Partial early virologic response | 5 | 0
  No early virologic response response | 10 | 14

4. Secondary Outcome: End-of-treatment Response
Description: An end-of-treatment response is defined as a negative HCV PCR at 48 weeks after the start of pegylated interferon and ribavirin
Time Frame: 48 weeks +- 7 days after starting pegylated interferon and ribavirin
Population: ITT. Any patient who received at least one dose of interferon was included in the analyses.
Measure: Number; unit: participants
Arm/Group | Standard of Care | Triple Therapy
Number analyzed (Participants) | 50 | 50
participants | 31 | 29

5. Secondary Outcome: Safety of Nitazoxanide (Number of Participants Experiencing Adverse Events)
Description: The occurence of adverse events that could be linked temporally and reasonably to the administration of the tested drug.
Time Frame: throughout the period of treatment and up to 90 days after end of triple therapy
Measure: Number; unit: participants
Arm/Group | Standard of Care | Triple Therapy
Number analyzed (Participants) | 50 | 50
participants | 50 | 47

ADVERSE EVENTS:
Arm/Group | Standard of Care | Triple Therapy
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 50/50 | 47/50
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=50) | Triple Therapy (N=50)
Fever (General disorders) | 49 | 45
Fatigue (General disorders) | 45 | 42
dyspepsia (Gastrointestinal disorders) | 7 | 16
anorexia (Gastrointestinal disorders) | 13 | 16
constipation (Gastrointestinal disorders) | 4 | 5
diarrhea (Gastrointestinal disorders) | 1 | 1
musculoskeletal pains (Musculoskeletal and connective tissue disorders) | 20 | 25
itching (Skin and subcutaneous tissue disorders) | 15 | 16
rash (Skin and subcutaneous tissue disorders) | 0 | 2
depression (Psychiatric disorders) | 4 | 4
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 6 | 2
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4
insomnia (Psychiatric disorders) | 5 | 2
headache (General disorders) | 16 | 24
Neutropenia (<1000/ml) (Blood and lymphatic system disorders) | 11 | 6
Anemia (Hgb <10g/dl) (Blood and lymphatic system disorders) | 16 | 15
facial palsy (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes